CLINICAL TRIAL: NCT01612819
Title: Evaluation of Effectiveness and Safety of DXR(Previous Cilotax) Stent in Routine Clinical Practice; A Multicenter Prospective Observational Cohort Study (IRIS-CILOTAX)
Brief Title: DXR Stent(Previous Cilotax) Implantation Registry
Status: Terminated | Type: Observational
Why Stopped: No more enrollment
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Cardiotec Corporation (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD, PhD, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: CVRF2012-01
Record Dates: First submitted 2012-06-01; First posted 2012-06-06 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Diseases
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Registry of cilotax stent(Dual drug eluting stent) implantation for CAD patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant coronary artery disease and receiving Cilotax (dual drug eluting stent)
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site

Exclusion Criteria:

* Patients with a mixture of other DESs
* Terminal illness with life expectancy <1 year
* Patients presented with cardiogenic shock

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery disease requiring drug eluting stents
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
composite of death, nonfatal myocardial infarction (MI), or target- Vessel Revascularization (TVR) | at 12 months post procedure

SECONDARY OUTCOMES:
Death (all cause and cardiac) | one month
Death (all cause and cardiac) | 6 months
Death (all cause and cardiac) | 12 months and yearly up to 5 years
Myocardial Infarction | 12 months and yearly up to 5 years
Myocardial Infarction | one month
Myocardial Infarction | 6 months
Composite of death or MI | 6 months
Composite of death or MI | one month
Composite of death or MI | 12 months and yearly upto 5 years
Composite of cardiac death or MI | one month
Composite of cardiac death or MI | 6 months
Composite of cardiac death or MI | 12 months and yearly up to 5 years
Target Vessel Revascularization | 12 months and yearly up to 5 years
Target Vessel Revascularization | one month
Target Vessel Revascularization | 6 months
Target-lesion revascularization | one month
Target-lesion revascularization | 6 months
Target-lesion revascularization | 12 months and yearly up to 5 years
Stent thrombosis | 12 months and yearly up to 5 years
Stent thrombosis | one month
Stent thrombosis | 6 months
Procedural success | at day 1
  It is defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Bae Seung, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital, Catholic University of Korea; Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (18):
- South Korea (18):
  - Soonchunhyang University Hospital, Buchen, Bucheon-si
  - Dankook University Hospital, Cheonan
  - Kangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daejeon St. Mary's Hospital, The Catholic University of Korea, Daejeon
  - GangNeung Asan Hospital, Gangneung
  - Gwangju Veterans Hospital, Gwangju
  - Kwangju Christian Hospital, Gwangju
  - Dongguk university gyeongju hospital, Gyeongju
  - Hallym University Dongtan Sacred Heart Hospital, Hwasŏng
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - ST.Carollo Hospital, Suncheon
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.